CLINICAL TRIAL: NCT05713266
Title: AIDI - Research and Development of a Multisensor-Based Technology for Real-time Automated Detection of Post-acute COVID-19 Sequelae
Brief Title: Using Data From a Multisensor Rapid Health Assessment Device to Predict Decompensation in Long COVID (AIDI)
Acronym: AIDI
Status: Completed | Type: Observational
Sponsor: Edith Nourse Rogers Memorial Veterans Hospital (U.S. Federal Agency)
Collaborators: AIDAR Health, Inc. (Industry); Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Principal Investigator, Varsha Vimalananda, MD, MPH, Physician-Scientist, Edith Nourse Rogers Memorial Veterans Hospital
Other Study IDs: 1720661-2
Record Dates: First submitted 2023-02-02; First posted 2023-02-06 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: COVID-19; Long COVID
Keywords: COVID-19; decompensation; long COVID-19; device; chronic kidney disease; diabetes; hypertension; asthma; chronic obstructive pulmonary diseaes; heart failure
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome; Renal Insufficiency, Chronic; Diabetes Mellitus; Hypertension; Asthma; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Severe COVID-19 survivors: Adult COVID-19 survivors who had 'severe COVID-19' during the acute phase and have at least one of the following pre-existing conditions: Hypertension, Asthma, COPD, Heart Failure, Chronic kidney disease and/or Diabetes. 'Severe COVID-19' is defined as requiring hospital or intensive level care for treatment of the infection and its complications.
  Interventions: Device: MouthLabTM

INTERVENTIONS:
Device: MouthLabTM — Aidar Health's MouthLab device is a non-invasive, hand-held, home monitoring tool that measures multiple clinically meaningful parameters such as temperature, blood pressure, heart rate, heart rate variability, pulse rate, SpO2, single-lead ECG, respiratory rate, breathing pattern, and basic lung functions in 60 seconds.

SUMMARY:
We are conducting a research study at the VA hospital in Bedford, MA to learn more about how a multisensor rapid health assessment device, MouthLab, can help predict or anticipate future health complications in patients with underline conditions after contracting COVID-19. The device was created by a health technology and digital medicine company called Aidar Health, Inc. MouthLab is a non-invasive, hand-held device that works like a breathalyzer. An individual breathes into the device for 60 seconds and the MouthLab gathers more than 10 vital health parameters like temperature, heart rate, SpO2, ECG, and basic lung functions. Participation in the study will last for 6 months, and the purpose is to gather health information from people who have been previously hospitalized with COVID-19. We will use the data to develop an algorithm that predicts future complications of COVID-19, especially among patients with complex conditions (i.e., heart failure, chronic kidney disease, diabetes, hypertension, asthma, chronic obstructive pulmonary disease), and enables early intervention.

DETAILED DESCRIPTION:
Severe complications like post-acute thrombosis, respiratory failure, and cardiac and vascular damage may increase the likelihood of future morbidity and mortality in recovered COVID-19 patients. Although the current rate of new COVID-19 infection has dropped, the risk of morbidity, mortality, and organ dysfunction among the survivors of COVID-19 infection is significant. An association between COVID-19 and an increased odds of acute kidney injury, renal replacement treatment, use of insulin, pulmonary embolism, stroke, myocarditis, arrhythmia, and increased troponin was found in US veterans admitted to hospital with COVID-19 versus a control group of patients with seasonal influenza. This comparative approach to examining post-acute sequelae in individuals who are hospitalized with COVID-19 versus individuals with seasonal influenza (using a high-dimensional approach and thorough examination of prespecified outcomes) suggests that there is a substantially higher burden of a broad array of post-acute sequelae in the individuals who are hospitalized with COVID-19, which provides features that differentiate post-acute COVID-19 (both in the magnitude of risk and the breadth of organ involvement) from a post-influenza viral syndrome.

Given the prevalence rates, it is evident that individuals in the post-acute phase even 12-months after their initial diagnosis continue to have abnormal physiological characteristics and increased utilization of healthcare resources as a consequence of altered health. This forces the conclusion that COVID-19 needs to be treated as a 'chronic condition' exhibiting an increased risk of morbidity, use of healthcare resources as well as a substantial burden of health loss that spans across pulmonary and extrapulmonary organ systems. From evidence and reasoning, it would be appropriate to infer that the next wave related to COVID-19 may not necessarily be a new strain but rather the surge of hospitalizations due to post-acute complications. Therefore, developing holistic and multidisciplinary long-term care strategies for patients with COVID-19 is emerging as an unmet need. To address these knowledge gaps, this study aims to recruit 'severe COVID-19' cases (i.e. those who required hospitalization during the acute COVID-19 phase), who have increased rates of multiorgan failure compared with the expected risk in the general population, to characterize the changes in cardiorespiratory parameters leading up to a decompensation event. Early prediction, real-time risk triaging shall be invaluable for better clinical decision making, preventing complications, controlling disease progression and improving outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Individuals who have had a COVID-19 related hospitalization (3-6 months prior to enrollment)
* Has at least one specified comorbidity (Diabetes, Heart Failure, Hypertension, Chronic Kidney Disease, Asthma, or COPD)
* Willing and able to provide informed consent
* Has no functional limitation that would impede the use of the MouthLab device, and is able to use the device with the left hand
* Comfortable with using technology
* Can commit to performing the required study tasks
* Can speak/understand English

Exclusion Criteria:

* Currently receiving hospice care
* Left-sided hemiplegia or any other motor deficits that may restrict the use of the device.
* Individuals with cognitive deficits that impede their ability to comprehend and give informed consent.
* Chest, abdominal or eye surgery within the preceding 14 days
* Any condition that in the judgment of the investigators would interfere with the subject's ability to provide informed consent, comply with study instructions, place the subject at increased risk, or which might confound interpretation of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who have tested positive for SARS-CoV-2 and required COVID-19 related hospitalization during the acute phase.
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2022-10-31 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
All cause higher level of care utilization | 6 months
  All cause higher level of care healthcare utilization (hospitalization, ER, or urgent care visits within VA system)

SECONDARY OUTCOMES:
All new diagnoses, treatment, utilization, medication | 6 months
  All new diagnoses, treatment, utilization, medication
Highly likely COVID-19 related diagnoses, treatment, utilization, medication | 6 months
  Highly likely COVID-19 related diagnoses, treatment, utilization, medication
Survey data | baseline, monthly and end of studu
  • Survey data
  * Self-reported presence of the following outcomes: (once a month)
    * MRC Dyspnea Scale (Score 1-5)
    * Post COVID-19 functional status scale (0-4 grade scale)
  * VR-12 Quality of Life Assessment (before and after the study)
  * MouthLab Usability Survey (Only after the study)
  * User Feedback on Remote Physiological Monitoring (RPM) technology
All cause healthcare utilization (within and outside VA) | 6 months
  All cause healthcare utilization (within and outside VA)
Highly likely COVID-19 related healthcare utilization | 6 months
  Highly likely COVID-19 related healthcare utilization
Highly likely+somewhat likely COVID-19 related healthcare utilization | 6 months
  Highly likely+somewhat likely COVID-19 related healthcare utilization

CONTACTS AND LOCATIONS:
Overall Officials: Varsha G Vimalananda, MD, MPH, Principal Investigator — Edith Nourse Rogers Memorial Veterans Hospital
Locations (1):
- VA Bedford Medical Center, Bedford, Massachusetts, United States

REFERENCES:
- [Derived] Pagliaro JA, Wash LK, Ly K, Mathew J, Leibowitz A, Cabrera R, Wormwood JB, Vimalananda VG. Enrollment and Retention Outcomes from the Veterans Health Administration for a Remote Digital Health Study: Multisite Observational Study. JMIR Form Res. 2025 Aug 15;9:e68676. doi: 10.2196/68676. PMID 40334212

DOCUMENTS (1):
  • Informed Consent Form (2023-02-16): https://cdn.clinicaltrials.gov/large-docs/66/NCT05713266/ICF_000.pdf